CLINICAL TRIAL: NCT03882541
Title: Could Music be an Alternative to Sedation in Patients Treated Total Knee Arthroplasty With Regional Anesthesia?: A Randomized Clinical Trial
Brief Title: Could Music be an Alternative to Sedation in Patients Treated Total Knee Arthroplasty With Regional Anesthesia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Anoia (Other)
Responsible Party: Principal Investigator, Sílvia Roca, Nurse, Consorci Sanitari de l'Anoia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRCSA0077
Record Dates: First submitted 2018-11-28; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2017-01

CONDITIONS: Anxiety; Surgery; Drug Toxicity; Anesthesia; Pain
Keywords: Anxiety; Pain; perioperative; Surgery; Music Therapy; Drugs
MeSH Terms: conditions — Anxiety Disorders; Drug-Related Side Effects and Adverse Reactions; Pain | interventions — Music Therapy; Midazolam

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): headphones without music, without sedation
- sedative group (Active Comparator): headphones without music, with sedation
  Interventions: Drug: Sedation with midazolam
- experimental group (Experimental): headphones with music, without sedation
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — To evaluate the effect of music in patients anxiety and pain during perioperative process in surgical intervention with regional anaesthesia without sedatives or anxiolytics.
  Arms: experimental group
Drug: Sedation with midazolam — To evaluate the effect of sedation (in comparation with music group) in patients anxiety and pain durin perioperative process in surgical intervention with regional anesthesia without music
  Arms: sedative group

SUMMARY:
Background: Anxiety is a common phenomenon in hospitalized patients. In order to reduce it during the surgical procedure, sedatives and anxiolytics are used, which can cause undesirable side effects for patients. Music is described as an effective tool to reduce this anxiety suffered by the patient in the perioperative process.

Objectives: To evaluate the effect of music in patients anxiety and pain during perioperative process in surgical intervention with regional anaesthesia without sedatives or anxiolytics.

Design: A randomized parallel clinical trial study with single-blinded and three harms.

Setting: Operating theater of a public district hospital (serving around 111.000 people) Participants: All patients operated of Total Knee Arthroplasty (TKA) with regional anaesthesia with age between 50 and 85 years old within level I or II of the classification of the American Society of Anaesthesiologists (ASA).

Methods: A total of 81 patients for TKA were randomly assigned to: a control group (headphones without music, without sedation), a sedative group (headphones without music, with sedation) and a experimental group (headphones with music, without sedation). 27 participants for each group. All the participants were using headphones so that it was a single-blinded study. The experimental group were provided with the same music, Piano Guys group. The variables of study were: the pain was measured by vale numerical scale (VNS), the anxiety was measured by the use of State-Trait Anxiety Inventory (STAI), heart rate (HR) variability, blood pressure (BP) variability, saturation of oxygen (Sat02).

Relevance to Clinical Practice: sedation that can causes unwanted side effects by surgical patients can be replaced by music. The music decrease anxiety and pain values in orthopaedic surgery patients.

Keywords: Anxiety, Drugs, Music therapy, Pain, Perioperative, Surgery.

DETAILED DESCRIPTION:
1. Introduction Patients generally experience high levels of anxiety when are hospitalized to undergo surgery and other invasive procedures. Anxiety is an emotional state or condition characterized by stress and unpleasant feelings. Awake patients in the operating theatre are afraid of they will feel pain during the surgical and/or regional anaesthetic procedures, which contributes to increased anxiety. Patients operated under regional anaesthesia are in particular need of sedation during the perioperative period. The purpose of the sedation is to ensure comfort, full cooperation and cardiovascular stability of patients who can maintain a patent airway. However, because of the adverse effects (respiratory depression, nausea, vomiting), optimal patient satisfaction is hard to achieve. Additionally, intraoperative anxiety is often associated with a greater incidence of pain after surgery.

   On the other hand, toxicity of general anaesthetics has been recently studied from its neurotoxic effect to neuroapoptosis. In some cases, they may cause postoperative cognitive dysfunction, and other side effects known as hypoxemia, respiratory depression and increased morbidity and mortality.

   Music has been suggested as a potential intervention to reduce anxiety and pain in the operating room environment. Systematic meta-analysis conducted by Nilsson revealed that 50% of studies (12 of 24) published between January 1995-January 2007 found significant reductions in anxiety scores as measured by STAI. and then more studies have been carried out on the benefits of music, which have continued to show that music reduces preoperative and postoperative anxiety and also reduces postoperative pain.

   There are also studies that conclude that patients to listening music require less midazolam to achieve a similar degree of relaxation as controls in ambulatory surgery patients and that the relaxing music a useful alternative to midazolam for pre-medication before surgery.

   Music holds considerable promise as an adjuvant pain management therapy and in mild cases may be used to supplement, perhaps even replace, pharmaceutical interventions before, during, and after painful procedures. The maximal reduction in pain intensity levels is 0.9 units on a zero to ten scale; although this difference reaches statistical significance, its clinical importance is unclear.

   The aim of this study was to evaluate the effect of the use of music in the perioperative process of patients undergoing surgery of total knee arthroplasty with regional anaesthesia without sedatives and compare anxiety and pain of these patients operated with regional anaesthesia, listening to or not music through headphones in patients without sedation.
2. Material and methods 2.1 Research design and setting This study was a randomized clinical trial study with single-blind, three harms and parallel, that took place in the operating theatre conducted from January 2017 to January 2018.

The participants who had the signed informed consent, once they reached the surgical area, were divided into the three groups according to the randomization list, control group (headphones without music, without sedation), sedation group (headphones without music, with sedation), intervention group (headphones with music, without sedation).

Ninety-five patients were eligible for the purpose of this study and ten were refused to participate in the study. From the 85 remaining subjects, 29 were allocated to the control group, 27 to the sedation group, while 29 were allocated to the intervention group. The CONSORT flow diagram of the progress through the phases of a parallel randomised trial of the three groups is shown on Figure 1.

There were not changes to methods after trial commencement.

2.2 Participants and Sample size The study was performed on participants scheduled for a Total Knee Arthroplasty procedure in a Public Hospital from January 2017 to January 2018. The inclusion criteria were: (1) age with a range from 50 to 85 years old, (2) had regional anaesthesia, (3) duration of surgery not exceeding two hours (4) was willing to participate in the study and signed an informed consent form. The exclusion criteria were: (1) those patients with classification system of American Society of Anaesthesiologists (ASA) 3 or 4, (2) allergic drugs used, (3) psychiatric patients or cognitive issues, (4) patients with whom we have communication problems, (5) patients who for any reason need another type of anaesthesia.

Sample size was determinate regarding the possible differences in the value of numerical pain among the 3 groups studied. Thus, in an analysis of the variance of a three-level factor (ANOVA), assuming a common standard deviation of 1.5 and a minimum difference to detect of 1 point (or equivalent, to detect a difference in any quantitative variable of 0,66 standard deviations), with a statistical power of 80% and an alpha error of 0.05, 53 patients were needed in each of the three groups to detect the difference as statistically significant. A maximum 10% follow-up loss was considered. The result of the sample was 159 participants. An interim analysis was carried out that according to the statistical calculation had to be carried out when arriving at 81 participants (27 for each group). If the result was significant beneficial or harmful compared to the concurrent placebo group the study could be stopped.

2.3 Randomization Randomization lists were generated based on pseudorandom numbers with the SPSS program. For the study, 3 blocks of 81 patients each were performed, corresponding to 27 patients for each group.

All randomization was independent of the researches. Randomization was done by a statistician who was not part of the data analysis.

When a participant was a candidate to participate in the study, the random allocation table was consulted when the group was assigned, the researchers elaborated a closed envelope with information on the intervention received (with or without sedation and with or without music) by the participant in case it was It is necessary to break the simple blind. They were also told to the participants that they would not say whether or not they would listen to music.

The staff, personnel and the assistants to the investigation were blinded to the participants group assignment.

2.4 Intervention Once the participants were included in the study, they were assigned a group according to the randomization table. The participants of the control group were placed with headphones that no produced music and were administered 2 ml of serum, participants in the sedation group were placed with headphones without music and were administered the corresponding dose of midazolam (0.025 mg / kg in patients under 65 years of age. In patients over 65 years of age and / or with hepatic insufficiency or renal insufficiency with glomerular filtration <30 ml / h, the dose of midazolam was 0.015 mg / Kg.) and the participants of the intervention group were placed with headphones that produced music and were administered 2 ml of serum. All the participants were administered the same anaesthetic (levobupivacaine) for regional anaesthesia and the same analgesics in the postoperative period (ropivacaine, dexketeroprofen, paracetamol). A standardization of anaesthesia and analgesia was performed by the anaesthesiology and resuscitation service of the hospital.

The music that the group's patients listened to during their stay in the operating theatre was a collection of songs from the music group Piano Guys, played a volume of 50-55 db. The headphone used were Audio-Technica ATH-M40X and the mp3 was iPod Nano (Apple).

According to some studies, it is recommended that therapeutic music should have a slow tempo, low pitch, regular rhythm, and pleasing harmonics, and should consist of string, flute, and piano selections (Nilsson, 2008; Pelletier, 2004). In a Cochrane review, the genre and the duration of the soothing music did not seem to influence the effectiveness of music intervention.

There were not any changes to trial outcomes after the trial commenced.

2.5 Instruments and Measurements We employed both subjective and objective measures for anxiety and pain in our study.

2.5.1 State-Trait Anxiety Inventory (STAI) The State-Trait Anxiety Inventory (STAI) consists of two different parts, termed STAI-Trait Anxiety Inventory (STAI-TA) and STAI-State Anxiety Inventory (STAI-SA). This test requires patients to complete a 40-item, 20 items measuring state anxiety and 20 items measuring trait anxiety (Spielberger et al.,1970) adding each one of the items of each subscale. The score can range between 0 and 60, representing the highest and lowest levels of anxiety, respectively. In our study, STAI-TA test results were evaluated preoperatively. The STAI-SA was performed during the waiting room (Orthopaedic unit, 30 minutes before surgery) and postoperative period in Post anaesthesia care unit (PACU) (recovery period, 30 minutes after surgery). There are no cut points, but direct scores are transformed into centiles based on sex and age.

2.5.2 Vale Numerical Scale (VNS) Pain intensity is frequently measured for visual analogue scale (VAS) or numerical ranting scale (NRS). We used the NRS, pain was assessed on a 10-point pain intensity numerical rating scale, where 0=no pain and 10=worst possible pain (Lee et al.2015). The researcher gave oral instruction of ''Please said the point at the number to show how much pain do you have right now''. The pain was measured in preoperative, intraoperative and postoperative phase.

2.5.3 Hemodynamic constants: To measure HR and BP, the researchers placed the sensor on the radial area of the patient's forearm for 15 minutes. Monitoring of the electrocardiogram (ECG) and capillary oxygen saturation (SatO2) was continuous. The participants were asked not to move around to ensure the quality of the readings. In our study, HR, BP and SatO2 was measured by a Datex Ohmeda TYPE D-LCC15..03.

2.6 Data collection process This research was approved by the Ethical Committee for Clinical Research, (approved code: PR218/16).

The researchers (SR, MR) checked the operating schedule and met potential participants in the room of orthopaedic unit where we take the signed consent and we gave them the STAI questionnaire.

When the participants reached preoperative area, the researchers looked the group that belonged to each participant according to randomization list and they were monitored hemodynamic constants (HR, BP, SatO2), the headphones were placed with or without music and the dose of sedation or physiological serum (placebo) was administrated according to the study group to which they belonged. The dose of sedation or serum was repeated every 45 minutes until surgery was finished. All the data (STAI preoperative and postoperative, VNS preoperative and postoperative, hemodynamic constants every 15 minutes, dose anaesthetics and analgesics, sociodemographic variables) were registered in a graph created by researchers.

The data collection in each phase, preoperative, intraoperative and postoperative, was carried out by nurses who did not belong to the research team, who were educated before starting the study so that there were no biases in the collection.

2.7 Statistical analysis Categorical variables were described by means of the number of cases, the percentage with respect to the total by category and the number of available data. Continuous variables were described by means of the number of cases, the mean and the standard deviation or the median and the inter-quartile range (IQR). Continuous variables were compared using Student's t-test or Mann-Whitney U-test as appropriate. Fisher's exact test or Pearson's χ2 test were applied to assess the relationship between categorical variables. In order to evaluate the main objective, a covariance analysis was performed to evaluate the role of the intervention in the change in the value of the final pain compared to initial pain. The effects of each intervention were compared by pairs with the adjustment for multiple comparisons of Tukey. The rest of the study variables (STAI questionnaire and hemodynamic constants (BP, HR, SatO2)) were analysed similarly. Models were replicated adjusted by age and gender. Analyses were performed with R software 3.4.0. The statistical significance was set at a probability level <0.05.

2.8 Ethical considerations The participants who met the inclusion criteria were informed by the researchers and they were also given an informative document of the study. The participants who wanted to participate in the study signed an informed consent.

4.1 Limitations When we performed the post-STAI test in the Post Anesthesia Care Unit (PACU), some patients could not read the questionnaire because they did not have the glasses, so the nurse had to ask the questions. In future studies, a better research design or a more suitable testing location can provide a better understanding on this subject. Additional research could examine the effectiveness of listening to preferred music, the use of music as an alternative to another type of sedative drug such as propofol, for other surgical patients, as well as their satisfaction.

Conflict of interest and Funding None Acknowledgements The authors thanks all professionals who have collaborated in the study: surgery nurses, nursing traumatology department and nursing supervision.

Thanks especially Dr Xavier Pelfort and Dr Joan Miquel, for assistance with study design, statistical analysis, manuscript review and anaesthetist Dr Josep Mª Bausili for assistance with anaesthesia standardization.

ELIGIBILITY:
Inclusion Criteria:

* Age with range from 50-85 years old
* Had regional anaesthesia
* Duration of surgery not exceeding two hours
* Was willing to participate in the study and signed an informed consent form

Exclusion Criteria:

* Those patients with classification system of American Society of Anaesthesiologist (ASA) 3 or 4
* Allergic drugs used
* Psychiatric patients or cognitive issues

  * Patients with whom we have communication problems
* Patients who for any reason need another type of anaesthesia.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-01-08 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Anxiety State-Trait Anxiety Inventory (STAI) | 10 minutes
  The State-Trait Anxiety Inventory (STAI) consists of two different parts, termed STAI-Trait Anxiety Inventory (STAI-TA) and STAI-State Anxiety Inventory (STAI-SA). This test requires patients to complete a 40-item, 20 items measuring state anxiety and 20 items measuring trait anxiety (Spielberger et al.,1970) adding each one of the items of each subscale. The score can range between 0 and 60, representing the highest and lowest levels of anxiety, respectively. In our study, STAI-TA test results were evaluated preoperatively. The STAI-SA was performed during the waiting room (Orthopaedic unit, 30 minutes before surgery) and postoperative period in Post anaesthesia care unit (PACU) (recovery period, 30 minutes after surgery). There are no cut points, but direct scores are transformed into centiles based on sex and age.

SECONDARY OUTCOMES:
Pain Vale Numerical Scale (VNS) | 3 minutes
  Pain intensity is frequently measured for visual analogue scale (VAS) or numerical ranting scale (NRS). We used the NRS, pain was assessed on a 10-point pain intensity numerical rating scale, where 0=no pain and 10=worst possible pain

OTHER OUTCOMES:
Heart Rate (pulsation for minute) | 15 minutes for 1 hour
  To measure HR, the researchers monitoring of the patient's with the electrocardiogram (ECG) and the monitoring was continuous.was measured by a Datex Ohmeda TYPE D-LCC15..03.
Blood Preasure (mmHg) | 15 minutes for 1 hour
  To measure BP, the researchers placed the sensor on the radial area of the patient's for arm for 15 minutes.was measured by a Datex Ohmeda TYPE D-LCC15..03.
Oxygen Saturation (%) | 15 minutes for 1 hour
  To measure oxygen saturation, the researches placed the sensor on the finger and this monitoring was continuous.was measured by a Datex Ohmeda TYPE D-LCC15..03.
Age (Years) | 1 minute
  in years
Gender (Male or Female) | 1 minute
  Male or female
Weight (in Kilogram) | 1 minute
  in kilogram

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allred KD, Byers JF, Sole ML. The effect of music on postoperative pain and anxiety. Pain Manag Nurs. 2010 Mar;11(1):15-25. doi: 10.1016/j.pmn.2008.12.002. Epub 2009 Mar 18. PMID 20207324
- [Background] Beccaloni AM. The medicine of music: a systematic approach for adoption into perianesthesia practice. J Perianesth Nurs. 2011 Oct;26(5):323-30. doi: 10.1016/j.jopan.2011.05.010. PMID 21939885
- [Background] Cepeda MS, Carr DB, Lau J, Alvarez H. Music for pain relief. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004843. doi: 10.1002/14651858.CD004843.pub2. PMID 16625614
- [Background] Cooke M, Chaboyer W, Schluter P, Hiratos M. The effect of music on preoperative anxiety in day surgery. J Adv Nurs. 2005 Oct;52(1):47-55. doi: 10.1111/j.1365-2648.2005.03563.x. PMID 16149980
- [Background] Good M, Anderson GC, Stanton-Hicks M, Grass JA, Makii M. Relaxation and music reduce pain after gynecologic surgery. Pain Manag Nurs. 2002 Jun;3(2):61-70. doi: 10.1053/jpmn.2002.123846. PMID 12050837
- [Background] Jimenez-Jimenez M, Garcia-Escalona A, Martin-Lopez A, De Vera-Vera R, De Haro J. Intraoperative stress and anxiety reduction with music therapy: a controlled randomized clinical trial of efficacy and safety. J Vasc Nurs. 2013 Sep;31(3):101-6. doi: 10.1016/j.jvn.2012.10.002. PMID 23953858
- [Background] Jevtovic-Todorovic V, Absalom AR, Blomgren K, Brambrink A, Crosby G, Culley DJ, Fiskum G, Giffard RG, Herold KF, Loepke AW, Ma D, Orser BA, Planel E, Slikker W Jr, Soriano SG, Stratmann G, Vutskits L, Xie Z, Hemmings HC Jr. Anaesthetic neurotoxicity and neuroplasticity: an expert group report and statement based on the BJA Salzburg Seminar. Br J Anaesth. 2013 Aug;111(2):143-51. doi: 10.1093/bja/aet177. Epub 2013 May 30. PMID 23722106
- [Background] Ilkkaya NK, Ustun FE, Sener EB, Kaya C, Ustun YB, Koksal E, Kocamanoglu IS, Ozkan F. The effects of music, white noise, and ambient noise on sedation and anxiety in patients under spinal anesthesia during surgery. J Perianesth Nurs. 2014 Oct;29(5):418-26. doi: 10.1016/j.jopan.2014.05.008. PMID 25261145
- [Background] Kushnir J, Friedman A, Ehrenfeld M, Kushnir T. Coping with preoperative anxiety in cesarean section: physiological, cognitive, and emotional effects of listening to favorite music. Birth. 2012 Jun;39(2):121-7. doi: 10.1111/j.1523-536X.2012.00532.x. Epub 2012 May 17. PMID 23281860
- [Background] Labrague LJ, McEnroe-Petitte DM. Influence of Music on Preoperative Anxiety and Physiologic Parameters in Women Undergoing Gynecologic Surgery. Clin Nurs Res. 2016 Apr;25(2):157-73. doi: 10.1177/1054773814544168. Epub 2014 Jul 30. PMID 25078946
- [Background] Lee JJ, Lee MK, Kim JE, Kim HZ, Park SH, Tae JH, Choi SS. Pain relief scale is more highly correlated with numerical rating scale than with visual analogue scale in chronic pain patients. Pain Physician. 2015 Mar-Apr;18(2):E195-200. PMID 25794219
- [Background] Lee KC, Chao YH, Yiin JJ, Chiang PY, Chao YF. Effectiveness of different music-playing devices for reducing preoperative anxiety: a clinical control study. Int J Nurs Stud. 2011 Oct;48(10):1180-7. doi: 10.1016/j.ijnurstu.2011.04.001. Epub 2011 May 11. PMID 21565344
- [Background] Lee KC, Chao YH, Yiin JJ, Hsieh HY, Dai WJ, Chao YF. Evidence that music listening reduces preoperative patients' anxiety. Biol Res Nurs. 2012 Jan;14(1):78-84. doi: 10.1177/1099800410396704. Epub 2011 Jan 28. PMID 21278165
- [Background] Ni CH, Tsai WH, Lee LM, Kao CC, Chen YC. Minimising preoperative anxiety with music for day surgery patients - a randomised clinical trial. J Clin Nurs. 2012 Mar;21(5-6):620-5. doi: 10.1111/j.1365-2702.2010.03466.x. Epub 2011 Feb 20. PMID 21332853
- [Background] Nilsson U. The anxiety- and pain-reducing effects of music interventions: a systematic review. AORN J. 2008 Apr;87(4):780-807. doi: 10.1016/j.aorn.2007.09.013. PMID 18395022
- [Background] Pelletier CL. The effect of music on decreasing arousal due to stress: a meta-analysis. J Music Ther. 2004 Fall;41(3):192-214. doi: 10.1093/jmt/41.3.192. PMID 15327345
- [Background] Shen X, Dong Y, Xu Z, Wang H, Miao C, Soriano SG, Sun D, Baxter MG, Zhang Y, Xie Z. Selective anesthesia-induced neuroinflammation in developing mouse brain and cognitive impairment. Anesthesiology. 2013 Mar;118(3):502-15. doi: 10.1097/ALN.0b013e3182834d77. PMID 23314110